CLINICAL TRIAL: NCT04560192
Title: Analysis of the Neuronal Correlates of a Mindfulness Based Emotion Regulation Therapy in the Treatment of Depressive Rumination Untersuchung Der Neuronalen Korrelate Eines Emotionsregulationstrainings Zur Behandlung Depressiven Grübelns
Brief Title: Mindfulness Based Emotion Regulation Therapy in the Treatment of Depressive Rumination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 159/2018BO1
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder; Depression; Rumination
Keywords: fNIRS; Rumination; Depression; Momentary Assessment; TSST; Emotion regulation therapy; Mindfulness based
MeSH Terms: conditions — Depressive Disorder; Depression; Rumination Syndrome | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Active Comparator): Treatment with the mindfulness based emotion regulation therapy (MBERT) in block 1, no study-treatment in block 2 (but patients receive their possibly already started treatment as usual including pharmacotherapy and psychotherapy).
  Interventions: Behavioral: Mindfulness based Emotion regulation therapy (MBERT) - Treatment as usual (TAU)
- Treatment as usual (TAU) (Other): No study-treatment in block 1 (but patients receive their possibly already started treatment as usual including pharmacotherapy and psychotherapy), treatment with the mindfulness based emotion regulation therapy (MBERT) in block 2.
  Interventions: Other: Treatment as usual (TAU) - Mindfulness based Emotion regulation therapy (MBERT)
- Control condition (No Intervention): Healthy subjects will get a single TSST session.

INTERVENTIONS:
Behavioral: Mindfulness based Emotion regulation therapy (MBERT) - Treatment as usual (TAU) — 1. In each of 8 sessions (allocated over 4 weeks) the patient brings an (actual) topic that induces rumination. After identifying the underlying affect, the patients are instructed (1) to concentrate on it, (2) to accept and tolerate it (considering the personal situation and experiences), (3) to give it a new interpretation so the patient can look at it with a more generous view, and (4) to dissociate from it, so the patient can perceive it as one of many affects and as one that hasn't the power to influence one's thoughts and actions that much (as it does through rumination). These steps are gradually instructed and trained throughout 20 trials (à 40 seconds) in each session. After each trial there is room to talk about the trial, possible barriers and helpful strategies to overcome those. Between-sessions the patients are encouraged to train the strategies in their daily life and do some homework like a protocol of ruminative thoughts and meditation.
  2. Waiting period with TAU.
  Arms: Intervention group
Other: Treatment as usual (TAU) - Mindfulness based Emotion regulation therapy (MBERT) — 1. Waiting period with TAU.
  2. In each of 8 sessions (allocated over 4 weeks) the patient brings an (actual) topic that induces rumination. After identifying the underlying affect, the patients are instructed (1) to concentrate on it, (2) to accept and tolerate it (considering the personal situation and experiences), (3) to give it a new interpretation so the patient can look at it with a more generous view, and (4) to dissociate from it, so the patient can perceive it as one of many affects and as one that hasn't the power to influence one's thoughts and actions that much (as it does through rumination). These steps are gradually instructed and trained throughout 20 trials (à 40 seconds) in each session. After each trial there is room to talk about the trial, possible barriers and helpful strategies to overcome those. Between-sessions the patients are encouraged to train the strategies in their daily life and do some homework like a protocol of ruminative thoughts and meditation.
  Arms: Treatment as usual (TAU)

SUMMARY:
In this study the investigators are examining the neuronal processes of a mindfulness based emotion regulation training for reducing depressive rumination. The research of depressive rumination helps in the developement of new therapies for depressive disorders.

Goal of this project is to have a look at the coherences between stress, mindfulness resources, depressive rumination and their neuronal correlates. Therefore the investigators are collecting the data of 48 patients with a depressive diagnosis in a randomized intervention-study with a treatment as usual (TAU) waiting-control-list versus an active intervention group. An additional 48 healthy control subjects are planned to be measured.

DETAILED DESCRIPTION:
In a randomized and (for gender and severity of depressive symptomatic) outbalanced design the investigators are examining the neuronal processes of a mindfulness based emotion regulation training (MBERT) for reducing depressive rumination in a cross-over design.

Therefore 48 patients with a depressive disorder get a MBERT that consists of one psychoeducative session and 8 therapy sessions.

For checking the efficacy of the MBERT each patient runs three times through the Trier Social Stress Test (TSST). As the study design is a cross-over design, half of the patients get the MBERT in block 1 (i.e. between the first and the second TSST) and half of the patients get the MBERT in block 2 (i.e. between the second and the third TSST). In the block where they don't receive the MBERT the patients don't get any treatment within the scope of the study (waiting period), but any treatment as usual (TAU), including pharmacotherapy and psychotherapy, can be continued and started at each point of the study.

For analyzing the neuronal processes the investigators are measuring the cerebral oxygenation using functional near-infrared-spectroscopy (fNIRS) during the TSSTs as well as during the 8 therapy sessions.

Using an ecological momentary assessment (EMA), the investigators additionally are collecting data of the actual stress level, stressful events, rumination, equanimity, self-compassion, mindfulness and sleep quality two times a day. Thus the investigators can (1) observe the individual reaction to stress in the daily life, and (2) recheck if the patients are able to transfer the learned strategies from the MBERT in their daily life. For those patients that received the MBERT in the first block the investigators (3) additionally have data to evaluate the sustainability (i.e. the lasting effectivity) of the MBERT.

As a control condition, 48 healthy subjects will get a single TSST session.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-60
* german as mother tongue
* diagnosis of a unipolar depressive disorder
* ruminative processes in the psychopathology

Exclusion Criteria:

* pregnancy
* acute or chronic disorder or medical treatment of such that might influence the cerebral metabolism:
* Diabetes mellitus (E10-E14 in ICD-10)
* Renal insufficiency apart from stadium 3 in Kidney Disease Outcomes Quality Initiative
* non adjusted hypertonus (I10.x in ICD-10)
* medium-severe or severe craniocerebral injury (GCS 3-12) / craniocerebral injury of 2. or 3. degree with loss of consciousness of > 30 minutes
* any medication except oral contraceptives
* other axis-I / axis-II disorders as main diagnosis
* comorbid neurological disease
* psychotic symptoms
* acute suicidality & very severe depressive symptomatology (BDI-II Score > 40)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-compassion-scale (SCS) | 8-10 weeks
  Changes in self compassion through the mindfulness based emotion regulation therapy. Minimum value: 1; maximum value: 5; higher values mean better self compassion (i.e. a better outcome).
Becks Depression Inventory (BDI) | 8-10 weeks
  Changes in depressive symptomatic through the mindfulness based emotion regulation therapy. Minimum value: 0; maximum value: 63; higher values mean more severe depressive symptoms (i.e. a worse outcome).
TSST | 3 times in 8-10 weeks
  Changes in behavior while and immediately after the stress induction via the Trier Social Stresstest
state rumination | 3 times in 8-10 weeks
  Changes in state rumination while and immediately after the stress induction via the Trier Social Stresstest; increase from pre to post TSST

SECONDARY OUTCOMES:
fNIRS TSST activation | 3 times in 8-10 weeks
  Hemodynamic response / brain activation while control tasks and the stress induction via the Trier Social Stresstest
fNIRS Training activation | 8 times in 4-5 weeks
  Hemodynamic response / brain activation while the mindfulness based emotion regulation therapy / training sessions
Training rating scores | 8 times in 4-5 weeks
  Friendliness (with oneself and ones emotions) as well as emotional distancing while the mindfulness based emotion regulation therapy / training sessions via single questions after each trial. Ratings range from 0 to 9, while the higher the score the more the friendliness or the emotional distancing (i.e. higher scores mean a better outcome).
Electronical momentary assessment (EMA) | 2 times per day in 8-10 weeks
  Self compassion, rumination, mindfulness, subjective stress and sleep quality in the daily routine (recorded via momentary assessment). Therefore items from different questionnaires (Self compassion scale (SCS), Ruminative Response Scale (RRS), Perseverative Cognitions Questionnaire (PCQ)) and self created items were taken. For self compassion, rumination and mindfulness mean scores can be calculated afterwards (self compassion: min: 0, max: 100; rumination & mindfulness: min: 0, max: 5; for self compassion and mindfulness higher scores mean a better outcome, for rumination higher scores mean a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Christine Ehlis, Dr., Study Chair — submitter and head of the lab
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Other researchers can get IPD of interest after request.
Supporting Information: Study Protocol
Time Frame: After publication
Access Criteria: Requester should have a scientistic (i.e. thematically related or complementary) interest in the data.

REFERENCES:
- [Derived] Laicher H, Int-Veen I, Woloszyn L, Wiegand A, Kroczek A, Sippel D, Leehr EJ, Lawyer G, Albasini F, Frischholz C, Mossner R, Nieratschker V, Rubel J, Fallgatter A, Ehlis AC, Rosenbaum D. In situ fNIRS measurements during cognitive behavioral emotion regulation training in rumination-focused therapy: A randomized-controlled trial. Neuroimage Clin. 2023;40:103525. doi: 10.1016/j.nicl.2023.103525. Epub 2023 Oct 13. PMID 37839195